CLINICAL TRIAL: NCT00518492
Title: Duration of Immunity in Healthy Adult Volunteers Who Completed Study 6108A1-500
Brief Title: Study Evaluating the Duration of Immunity in Healthy Adult Volunteers Who Completed Study 6108A1-500
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6108A1-1002
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Includes subjects from a trial involving experimental vaccine and an active comparator vaccine. Comparator is Twinrix (not a MnB vaccine) and thus is comparator for safety but not immunogencity
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — Blood draws at 6 and 12 months following end of 6108A1-500 trial.

SUMMARY:
Upon completion of participation in the 6108A1-500 study, subjects will be asked to consent for this duration of immunity study to provide up to two additional blood samples. SBA & IgG testing will be done on these samples taken at 6 & 12 months. The sites participating in this duration of immunity study are the same sites participating in the 6108A1-500 study.

ELIGIBILITY:
Inclusion Criteria:

* Completed study 6108A1-500 (three doses administered and visit 9 completed).

Exclusion Criteria:

* Bleeding diathesis or condition associated with prolonged bleeding time.
* Any clinically significant chronic disease that, in the investigators judgment may be worsened by blood draw.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity at 6 and 12 months post 6108A1-500 study. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia: medinfo@wyeth.com
Locations (3):
- Australia (3):
  - Herson, Queensland
  - North Adealaide, South Australia
  - Perth, Western Australia